CLINICAL TRIAL: NCT02083250
Title: Fludarabine/Clofarabine/Busulfan Combined With SAHA in Patients Receiving Allogeneic Hematopoietic Stem Cell Transplantation for Acute Leukemia
Brief Title: Fludarabine Phosphate, Clofarabine, and Busulfan With Vorinostat in Treating Patients With Acute Leukemia in Remission or Relapse Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0999; NCI-2014-01982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0999 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Clofarabine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vorinostat, chemotherapy, SCT) (Experimental): CONDITIONING REGIMEN: Patients receive vorinostat PO QD, fludarabine phosphate IV over 1 hour, clofarabine IV over 1 hour, and busulfan IV over 3 hours on days -6 to -3. Patients receiving a transplant from a HLA-matched unrelated donor, receive anti-thymocyte globulin IV over 4 hours on days -3 to -1.
  TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell or bone marrow transplant on day 0.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Clofarabine; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Vorinostat

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic peripheral blood stem cell or bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell or bone marrow transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell or bone marrow transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I trial studies the side effects and best dose of vorinostat when given together with fludarabine phosphate, clofarabine, and busulfan in treating patients with acute leukemia that is under control (remission) or has returned (relapse) undergoing donor stem cell transplant. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine phosphate, clofarabine, and busulfan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving vorinostat together with fludarabine phosphate, clofarabine, and busulfan before a donor stem cell transplant may be a better treatment for patients with acute leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of SAHA (vorinostat) in combination with the preparative regimen fludarabine (fludarabine phosphate), clofarabine, and busulfan followed by allogeneic hematopoietic stem cell transplantation (SCT) for patients with advanced acute leukemia.

SECONDARY OBJECTIVES:

I. To determine the rate of graft versus host disease (GVHD), engraftment, progression-free survival (PFS) and overall survival (OS) for this treatment regimen.

OUTLINE: This is a dose-escalation study of vorinostat.

CONDITIONING REGIMEN: Patients receive vorinostat orally (PO) once daily (QD), fludarabine phosphate intravenously (IV) over 1 hour, clofarabine IV over 1 hour, and busulfan IV over 3 hours on days -6 to -3. Patients receiving a transplant from a human leukocyte antigen (HLA)-matched unrelated donor, receive anti-thymocyte globulin IV over 4 hours on days -3 to -1.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell or bone marrow transplant on day 0.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven acute lymphoblastic leukemia, acute myeloid leukemia, or myelodysplastic syndrome in remission or relapse
* Estimated creatinine clearance at least 50 ml/min
* Bilirubin equal or less than 1.5 (unless Gilbert's syndrome)
* Serum glutamate pyruvate transaminase (SGPT) < 3 x upper limit of normal
* Alkaline phosphatase < 2 x upper limit of normal
* Pulmonary function with forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lungs for carbon monoxide (DLCO) at least 45% of expected corrected for hemoglobin; children unable to perform pulmonary functions must have an oxygen saturation greater than 92% at room air
* Left ventricular ejection fraction at least 45% on appropriate medical therapy; no uncontrolled arrhythmias or symptomatic cardiac disease
* Zubrod performance status 0-1 or Lansky/Karnofsky performance status (PS) equal or greater to 80%
* Patients must have a related, genotypically HLA identical donor, or they must have an unrelated donor who is 8/8 HLA match by high resolution typing
* Patient or patient's legal representative, parent(s) or guardian should provide written informed consent; assent of a minor if participant's age is at least seven and less than eighteen years
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months and no previous surgical sterilization

Exclusion Criteria:

* Patients with active central nervous system (CNS) disease
* Evidence of acute or chronic active hepatitis or cirrhosis
* Uncontrolled infection, including human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV)-1, hepatitis B or hepatitis C viremia
* Prior allogeneic SCT
* Prior autologous SCT in last 12 months
* Patients with acute myeloid leukemia (AML) in first remission after one course of induction and with favorable cytogenetics (t[8;21], inv 16, or t[15;17]) and/or molecular profile (nucleophosmin [NPM]1)
* Prior radiation to liver in form of total body or involved field

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat when given in combination with fludarabine phosphate, clofarabine, and busulfan before stem cell transplant assessed using Common Terminology Criteria for Adverse Events version 4 | 30 days
  The 2-stage time-to-event continual reassessment method will be used. Toxicity will be tabulated by dose, type, and grade. The probability of toxicity over 30 days as a function of dose will be estimated by fitting a Bayesian binary outcome regression model.

SECONDARY OUTCOMES:
Recurrence-free survival | Up to 5 years
  Will be estimated by the Kaplan and Meier method.
Overall survival | Up to 5 years
  Will be estimated by the Kaplan and Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org